CLINICAL TRIAL: NCT04919746
Title: Change in Dielectric Constant, Elasticity and Temperature by Stimulation of Systemic Acupuncture Points
Brief Title: Change in Dielectric Constant, Elasticity and Temperature by Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, Elaine Caldeira de Oliveira Guirro, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4749033/2021
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Acupuncture
Keywords: Acupuncture; Lower limb

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group Acupuncture 1 - GA1 (Experimental): Healthy individuals aged between 18 and 38 years. The dielectric constant will be evaluated with a depth measurement of 0.5 mm, elasticity and infrared thermography in the region of the systemic acupuncture points.
  Interventions: Other: Systemic acupuncture
- Group Acupuncture 2 - GA2 (Experimental): Healthy individuals aged between 18 and 38 years. The dielectric constant will be evaluated with a depth measurement of 2.5 mm, elasticity and infrared thermography in the region of the systemic acupuncture points.
  Interventions: Other: Systemic acupuncture
- Group Acupuncture 3 - GA3 (Experimental): Healthy individuals aged between 18 and 38 years. The dielectric constant will be evaluated with a depth measurement of 5.0 mm, elasticity and infrared thermography in the region of the systemic acupuncture points.
  Interventions: Other: Systemic acupuncture
- Group Control 1 - GC1 (No Intervention): Healthy individuals aged between 18 and 38 years. The dielectric constant will be evaluated with a depth measurement of 0.5 mm, elasticity and infrared thermography in the region of the systemic acupuncture points.
- Group Control 2 - GC2 (No Intervention): Healthy individuals aged between 18 and 38 years. The dielectric constant will be evaluated with a depth measurement of 2.5 mm, elasticity and infrared thermography in the region of the systemic acupuncture points.
- Group Control 3 - GC3 (No Intervention): Healthy individuals aged between 18 and 38 years. The dielectric constant will be evaluated with a depth measurement of 5.0 mm, elasticity and infrared thermography in the region of the systemic acupuncture points.

INTERVENTIONS:
Other: Systemic acupuncture — Systemic acupuncture will be performed on the lower limb, bilaterally, at points E36 (Zusanli) and BP6 (Sanyinjiao). Point location specificity will be determined using the anatomical and directional F-cun reference method. Stimulation of pre-defined points will be performed using needles with a threadlike, sterile, disposable character and size 0.25 x 30.0 mm, within a period of 20 minutes. The insertion of the needle will be at a depth of 0.5 inches, aiming to obtain the De Qi, sensation of energy at the point and in the corresponding meridian, referring to the effectiveness of systemic acupuncture.
  Arms: Group Acupuncture 1 - GA1; Group Acupuncture 2 - GA2; Group Acupuncture 3 - GA3

SUMMARY:
Evaluate the effect of systemic acupuncture on dielectric constant, elasticity and skin temperature in healthy individuals.

DETAILED DESCRIPTION:
Systemic acupuncture is a therapeutic resource in Chinese Medicine that uses needles at specific points in the body, consistent with a system called acupuncture meridians. The aim of the study is to evaluate the effect of systemic acupuncture on dielectric constant, elasticity and skin temperature in healthy individuals. Will be evaluated 360 volunteers aged between 18 and 38 years and both sexes divided into six homogeneous groups. Pregnant women or those with a delay in the menstrual cycle for more than 28 days will be excluded. The evaluation will consist of measuring the dielectric constant at different depths of the skin, elasticity and infrared thermography of systemic acupuncture points. The procedure will be performed in three moments: pre systemic acupuncture (prior to stimulation), immediate post-systemic acupuncture (20 minutes after the start of stimulation), and post systemic acupuncture (40 minutes after the start of stimulation). Systemic acupuncture will be performed on the lower limb, bilaterally, at points E36 (Zusanli) and BP6 (Sanyinjiao), lasting 20 minutes. The multiple comparison ANOVA test will be performed, with statistical significance of 5% (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged between 18 and 38 years, both genders and without health complaints.

Exclusion Criteria:

* Pregnant female volunteers or those with a delay in the menstrual cycle for more than 28 days.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-08-02 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Dielectric constant | 10 minutes
  MoistureMeterD
Elasticity | 10 minutes
  ElastiMeterD
Infrared thermography | 15 minutes
  FLIR Systems T300